CLINICAL TRIAL: NCT00229918
Title: Combined Posterior Sub-Tenon Injection of Triamcinolone Acetonide and Laser Photocoagulation for the Treatment of Clinically Significant Macular Edema
Brief Title: PST/Laser v. Laser Alone for CSME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PST/CSME
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2005-09-30 (Estimated); Status verified 2005-09

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic macular edema; Clinically significant macular edema
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: triamcinolone acetonide

SUMMARY:
Prospective randomized clinical trial comparing Laser Alone v. Laser and posterior sub-tenon injection of triamcinolone acetonide for primary and refractory clinically significant macular edema.

DETAILED DESCRIPTION:
Clinically significant macular edema (CSME) is one of the leading causes of vision loss in diabetic retinopathy. The current standard of care for CSME is focal/grid laser photocoagulation. However, many patients experience further vision loss and/or require multiple laser treatments. In recent studies, intraocular (intravitreal) injection of triamcinolone acetonide has been shown to be beneficial for CSME, however, risks of this procedure include endophthalmitis and increased risk of steroid-induced intraocular pressure (IOP) elevation. Posterior sub-Tenon injection (PST) of triamcinolone acetonide is commonly used for inflammatory conditions of the eye and recently, has been increasingly used for diabetic macular edema. The objective of this study is to determine whether combined treatment with PST triamcinolone acetonide and laser photocoagulation for CSME has decreased rates of moderate vision loss, increased visual gain, and decrease in central macular thickness compared to laser photocoagulation alone. Both primary (no previous history of focal/grid laser) and refractory (previous history of focal/grid laser) CMSE will be studied. Thirty (30) eyes with primary CSME and thirty (30) eyes with refractory CSME will be randomized into one of two groups: 1) PST/Laser group and 2) Laser alone group. All patients will have an Optical Coherence Tomography (OCT) at the initial and final visits. Patients assigned to PST/Laser group will use topical steroid (1% prednisolone acetate) four times a day for two weeks. Patients who have elevated IOP with topical steroids will not receive PST steroid injection. Following treatments, patients will be evaluated at 1 and 2 months for a dilated eye exam, visual acuity, and assessment of IOP. Moderate vision loss (loss of 15 ETDRS letters), vision gain (in ETDRS letters), and central macular thickness (measured by OCT) will be compared between groups. Multivariate analysis will also be used to compare outcomes from the two arms of the study.

ELIGIBILITY:
Inclusion Criteria:

The criteria listed below must be satisfied in order for the patient to be eligible for the study.

* Age 25 to 80, inclusive.
* Primary CSME: CSME secondary to diabetic retinopathy as defined by the ETDRS in one or both eyes with no previous history of focal/grid laser photocoagulation.
* Refractory CSME: CSME secondary to diabetic retinopathy as defined by the ETDRS in one or both eyes with at least one session of focal/grid laser photocoagulation. Additionally, the eye must have a central macular thickness of at least 300 μM (normal, 200 μM) as measured by OCT and vision loss from baseline.

  * All patients in the Hines VA Eye Clinic with suspicion of CSME will be referred to the Hines VA Retina Clinic where they will be evaluated by a Retina specialist (Dr. De Alba) and where the diagnosis of CSME will be confirmed by clinical examination and fluorescein angiography.

Exclusion Criteria:

If any of the exclusion criteria listed below is/are present, the patient will not be eligible for the study.

* Unwilling or unable to give consent.
* Unable to return for scheduled follow-up visits.
* No light perception, light perception, count fingers, or hand motion vision.
* History of glaucoma (any form).
* History of ocular hypertension.
* History of IOP elevation with ocular and/or systemic steroid treatment.
* Baseline IOP greater than 22 mmHg.
* All patients with IOP elevation greater than 22 mmHg following treatment with topical prednisolone acetate.
* All patients with IOP elevation greater than 5 mmHg from baseline measurement following treatment with topical Prednisolone acetate.
* Advanced proliferative diabetic retinopathy.
* History of retinal detachment in either eye.
* Any ocular disease (anterior or posterior segment) obstructing the view of the fundus (i.e., dense cataract, vitreous hemorrhage).
* History of PST or intravitreal triamcinolone acetonide injection in either eye six months prior to the study.
* History of 20/200 vision or worse from any cause in the fellow eye.
* Active inflammatory, infectious, or idiopathic keratitis.

Ages: 25 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-09; Study Completion 2006-09

PRIMARY OUTCOMES:
Vision loss
Vision gain
Central macular thickness

SECONDARY OUTCOMES:
Increased intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Felipe de Alba, MD, Principal Investigator — Edward Hines Jr. VAH; Anuradha Khanna, MD, Principal Investigator — Edward Hines Jr. VAH
Locations (1):
- Edward Hines Jr. VAH, Hines, Illinois, United States